CLINICAL TRIAL: NCT03234647
Title: First In Human Study of the Doraya Catheter for the Treatment of AHF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revamp Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Doraya FIH Study for AHF
Record Dates: First submitted 2017-07-19; First posted 2017-07-31 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2018-09

CONDITIONS: Acute Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AHF patients (Experimental): AHF patient treatment with the Doraya catheter
  Interventions: Device: Doraya catheter

INTERVENTIONS:
Device: Doraya catheter — Temporary deployment of the Doraya catheter in AHF patients.

SUMMARY:
Safety and performance evaluation of the Doraya catheter in patients admitted with AHF.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to evaluate the safety and performance of the Doraya catheter in patients admitted with AHF, presenting persistent volume over load and poor response to diuretic treatment.

ELIGIBILITY:
Inclusion Criteria:

* AHF subjects with poor diuretic response

Exclusion Criteria:

* AHF subjects with sufficient diuretic response

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Device or procedure related Serious Adverse Event (SAE) rate through 60 days | 60 days
  SAE as defined by ISO 14155

CONTACTS AND LOCATIONS:
Overall Officials: Tal Hasin, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (7):
- Belgium (2):
  - Onze-Lieve-Vrouwziekenhuis Aalst, Aalst
  - ZNA Middelheim, Antwerp
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
- Poland (3):
  - Śląski Uniwersytet Medyczny w Katowicach, Katowice
  - 4th Military, Wroclaw
  - University Hospital, Wroclaw

REFERENCES:
- [Derived] Zymlinski R, Biegus J, Vanderheyden M, Gajewski P, Dierckx R, Bartunek J, Ponikowski P. Safety, Feasibility of Controllable Decrease of Vena Cava Pressure by Doraya Catheter in Heart Failure. JACC Basic Transl Sci. 2023 Apr 24;8(4):394-402. doi: 10.1016/j.jacbts.2023.02.010. eCollection 2023 Apr. PMID 37138800